CLINICAL TRIAL: NCT06928506
Title: RECLAIM: Recovering From COVID-19 Lingering Symptoms Adaptive Integrative Medicine Trial - Effect of Hi-OxSR for the Treatment of Post COVID Condition (RECLAIM-HiOxSR)
Brief Title: Effect of Hi-OxSR for the Treatment of Post COVID Condition
Acronym: RECLAIM-HiOxSR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-6203-HiOxSR
Record Dates: First submitted 2025-04-11; First posted 2025-04-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Long COVID; Post COVID-19 Condition; Post Acute Sequelae of COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: RECLAIM is a Canada-wide phase ll/lll, prospective, adaptive randomized controlled platform trial that is intended to study various interventions for the treatment of long COVID. Participants in the Hi-OxSR sub-protocol will be randomized in a 1:1:1 ratio to one of 3 arms.
Who Masked: Participant
Masking Description: Participants are not be blinded to group allocation, and will know what group they are assigned to. Participants will be masked to the hypothesis of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Use of Hi-OxSR for 30 minutes twice a day at low oxygen flow (0.5-3 liters per minute) for 2 weeks.
  Interventions: Device: Hi-OxSR device
- Group 2 (Experimental): Use of Hi-OxSR for 30 minutes twice a day at low oxygen flow (0.5-3 liters per minute) for 4 weeks.
  Interventions: Device: Hi-OxSR device
- Group 3 (Active Comparator): Use of Hi-Ox for 30 minutes twice a day at high oxygen flow (5 liters per minute) for 2 weeks.
  Interventions: Device: Hi-Ox device

INTERVENTIONS:
Device: Hi-OxSR device — The Hi-OxSR device consists of the Hi-Ox mask connected to a portable oxygen concentrator, with added tubing serving as a reservoir for rebreathed exhaled breath.
  Arms: Group 1; Group 2
Device: Hi-Ox device — The Hi-Ox mask is connected to a portable oxygen concentrator.
  Arms: Group 3

SUMMARY:
The RECLAIM study platform will be used to explore whether the use of the Hi-OxSR device improves the symptoms of post covid cognitive dysfunction. Carbon dioxide (CO2) has been proposed as a potential treatment for persistent immune activation as there is evidence that CO2 has antioxidant, anti-inflammatory, and anti-cytokine effects. We conducted a pilot study assessing the open label use of re-breathing CO2 (using Hi-OxSR) twice a day for 14 days, for the treatment of post-COVID cognitive dysfunction. Significant improvements were found in multiple cognitive assessments using TestMyBrain cognitive tests and brain fog (MSNQ) and fatigue scores. This phase 2 clinical trial seeks to build on current findings to determine the optimal effective dose of treatment (i.e. length of use, oxygen concentration, without or without CO2 rebreathing) and the safety of using Hi-OxSR in this patient population.

DETAILED DESCRIPTION:
This is a Sub-Protocol to the Core Clinical Study Protocol titled: REcovering from COVID-19 Lingering symptoms Adaptive Integrative Medicine (RECLAIM)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Positive COVID-19 test by nasopharyngeal swab RT-PCR (reverse transcription polymerase chain reaction) test, antibody or antigen tests at least 3 months prior to randomization; OR Presumed COVID-19 assessed by the site investigator (no positive COVID-19 test) with acute illness after October 15, 2019.
3. Patients should be treated with standard of care therapies (as discussed in the study manual) for at least 4 weeks prior to entry into trial.
4. Lingering COVID-19 symptoms beyond 3 months from onset of acute COVID and symptoms have lasted at least 2 months. The onset of COVID is considered the earliest of two dates: the date of positive test or the date of first symptoms;
5. Lingering symptoms from COVID-19 present at the time of randomization. "Lingering symptoms of Long COVID" must include self-reported cognitive dysfunction symptoms.
6. Female patients of childbearing potential (as assessed by the overseeing Investigator) who are sexually active must agree to practice true abstinence or use effective methods of contraception while on study treatment. Effective methods of contraception must be discussed and approved by the overseeing Investigator.
7. Must be able to provide informed consent and both willing and able to comply with study requirements.
8. Oxygen saturation on room air ≥92% at screening measured by pulse oximeter.

Exclusion Criteria:

1. Patients who had mechanical ventilation or extracorporeal membrane oxygen (ECMO) for COVID-19;
2. Current end-organ failure, organ transplantation, or current hospitalization in acute care hospital;
3. Contraindications to all of the study interventions;
4. Co-enrolment in another interventional trial (co-enrolment in an observational study is permitted);
5. Currently pregnant or breastfeeding.
6. Known physician diagnosis of cognitive dysfunction prior to COVID infection
7. Use of an investigational drug/device or other interventions within 30 days of screening
8. Use of home oxygen (O2) at baseline
9. History of pulmonary hypertension
10. Interstitial pulmonary fibrosis
11. Moderate to severe chronic obstructive pulmonary disease (COPD)
12. History of narcolepsy
13. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the participant or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Simple reaction time (SRT) task from the TestMyBrain (TMB) Digital Neuropsychology Toolkit On-line survey tool | Baseline/Start of intervention to two months
  TestMyBrain was developed as a tool to collect large, population-based samples for understanding the relationship between cognition, emotion, social functioning, and health. This test will take about 5 minutes to complete and will assess reaction time.
Verbal paired associates (VPA) task from the TestMyBrain (TMB) Digital Neuropsychology Toolkit On-line survey tool | Baseline/Start of intervention to two months
  TestMyBrain was developed as a tool to collect large, population-based samples for understanding the relationship between cognition, emotion, social functioning, and health. This test will take about 5 minutes to complete and will assess memory.

SECONDARY OUTCOMES:
All cognitive performance tasks (measured by the TESTMYBRAIN.org (TMB) neuropsychology toolkit | Baseline/start of intervention to 2 weeks, 1, 2 and 6 months
  TestMyBrain was developed as a tool to collect large, population-based samples for understanding the relationship between cognition, emotion, social functioning, and health. This test battery will take about 20 minutes to complete and will assess: verbal, episodic and working memory, attention, processing speed, basic psychomotor response speed, and cognitive control.
Brain Fog Questionnaire | Baseline/start of intervention to 2 weeks, 1, 2 and 6 months
  (Adapted from MSNQ) This is a self-administered 15-item questionnaire that assesses neurocognitive function. It takes approximately less than 5 minutes to complete
Brief Fatigue Inventory | Baseline/start of intervention to 2 weeks, 1, 2 and 6 months
  The self-administered Brief Fatigue Inventory is composed of 9 items evaluated on a 10-point scale, assessing severity of fatigue and impact of fatigue on daily life. It takes approximately 2-3 minutes to complete.
Short Form (SF)-36 | Baseline/start of intervention to 2 weeks, 1, 2 and 6 months
  Mental health related quality of life, measured by the Mental Composite Score (MCS), and physical health-related quality of life, measured by the Physical Component Score (PCS) of the SF-36 (v.1)
Safety, adverse events and serious adverse events | Baseline/start of intervention to 6 months
  Safety of the Hi-OxSR device will be reported through Adverse Events (AEs) and Serious Adverse Events (SAEs) throughout the study period.
Symptom Checklist | Baseline/start of intervention to 2 and 6 months
  Symptom Checklist (adapted from the De Paul Symptom Questionnaire (DSQ2), the World Health Organization Global COVID-19 Clinical Platform's Post COVID-19 case report form (CRF) and the Symptom Burden Questionnaire for Long COVID): to track symptom trajectory.
The DePaul Symptom Post-Exertional Malaise Short Form DSQ-PEM | Baseline/start of intervention to 2 weeks, 1, 2 and 6 months
  The self-administered DSQ-PEM is comprised of two sections assessing post-exertional malaise (PEM): (i) frequency and severity of PEM (5 questions), (ii) consequences, symptoms and recovery (5 questions).
Dyspnea | Baseline/start of intervention to 2 and 6 months
  Assessed using the Borg Dyspnea scale. This short assessment tool assesses perceived shortness of breath on exertion using a 10 point scale as assessed by the patient.
Mental Health - General Anxiety Assessment Form (GAD-7) | Baseline/start of intervention to 2 and 6 months
  The GAD-7 is a valid and efficient tool for screening for generalized anxiety disorder and assessing its severity in clinical practice and research. It is an easy-to-use, self-administered patient questionnaire that can be completed in minutes.
Mental Health - Patient Health Questionnaire (PHQ-9) | Baseline/start of intervention to 2 and 6 months
  The PHQ-9 is a validated, multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It incorporates Diagnostic and Statistical Manual IV (DSM-IV) depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. The PHQ-9 is brief and useful in clinical practice.
Mental Health -Post-traumatic Stress Disorder Checklist (PCL-5) | Baseline/start of intervention to 2 and 6 months
  The PCL-5 is a validated, reliable, 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual 5 (DSM-5) symptoms of Post-Traumatic Stress Disorder (PTSD). It takes approximately 5-10 minutes to complete.
Reintegration to Normal Living Index (RNLI) | Baseline/start of intervention to 2 and 6 months
  This short self-administered assessment tool will determine the degree to which participants reintegrate into normal social activities such as recreation, mobility in the community and interaction in family and other relationships. This tool has been validated in community living adults with mobility limitations.
Blood samples | Baseline/start of intervention and 2 months
  Blood samples will be used in correlative studies using advanced multi-omic and machine learning methods to better understand our results so as to identify phenotypes that will benefit from specific therapies
Fatigue Scale (adapted from the De Paul Symptom Questionnaire (DSQ2) | Baseline/start of intervention to 2 weeks, 1, 2 and 6 months
  The Fatigue Scale was adapted from the De Paul Symptom Questionnaire (DSQ2)'s 38 questions assessing medical history of Myalgia encephalomyelitis/chronic fatigue syndrome (ME/CFS), comorbidities, medications, impact on quality of life and daily activities, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Cheung, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - University Health Network, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec